CLINICAL TRIAL: NCT06280690
Title: SGM-101 Tumor-targeted Fluorescence Endoscopy to Enable Discrimination of Malignant From Benign Tissue in Rectal Polyps With Suspected T1 Adenocarcinoma or High Grade Dysplasia: a Feasibility Study
Brief Title: SGM-101 Tumor Targeted Fluorescence Endoscopy in Rectal Polyps With Suspected T1 Adenocarcinoma or High Grade Dysplasia
Acronym: SGM-T1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Dr. A.L. Vahrmeijer, Leiden University Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NL83765.058.23
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer; Image; Low Grade Dysplasia of Colon
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single center prospective, non-randomized phase 2 proof of concept study, on the performance of SGM-101 to discriminate T1RC/HGD from LGD in patients that will be scheduled for endoscopic local en-bloc resection in the Leiden University Medical Centre (LUMC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10mg SGM-101 (Experimental): This cohort receives 10mg
  Interventions: Drug: SGM-101
- 5mg SGM-101 (Experimental): This cohort receives 5mg
  Interventions: Drug: SGM-101

INTERVENTIONS:
Drug: SGM-101 — SGM-101 is cea-targeted fluorescent dye

SUMMARY:
This will be the first trial investigating whether tumor targeted fluorescence is able to discriminate invasive T1 carcinoma / High grade dysplasia from Low grade dysplasia/normal tissue during endoscopic intraluminal resection. This will be done using the CEA-targeted fluorescent probe SGM-101.

DETAILED DESCRIPTION:
Selection of patients with early rectal cancer, T1 rectal cancer (T1RC) or high-grade dysplasia (HGD), for local resection is based on endoscopic imaging, endorectal ultrasound and/or MRI. However, all these imaging modalities have their limitations in the accurate detection of small areas of cancer in large rectal polyps. Fluorescent guided endoscopy may offer the opportunity to aid in detecting these small cancerous areas in colorectal polyps.

Detection of T1RC or HGD in large rectal polyps is essential to select patients for the appropriate (endoscopic) resection technique. Completely benign polyps, solely containing low-grade dysplasia (LGD), could be resected by piecemeal endoscopic mucosal resection (pEMR), a fast technique on which almost all endoscopists are trained. However, for rectal polyps with T1RC or HGD, curative resection must be achieved by en-bloc resection techniques such as endoscopic submucosal dissection (ESD) or endoscopic intermuscular dissection (EID). These techniques are more complex and expensive and only a small number of endoscopists are trained on these techniques. pEMR of lesions with HGD or T1RC must be avoided because they may result in irradical resections (R1) or in inconclusive histological margin assessment since the polyp is not resected en-bloc. Often, this leads to unnecessary additional abdominal surgical resections.

Furthermore reported sensitivities for optical diagnosis of T1RC in a polyp are low, varying from 20.8% to 77.8%. Because of the limited accuracy of optical diagnosis, the current Dutch guideline suggest that rectal polyps >3cm should be resected in an en-bloc manner, although it has been demonstrated that only 10.2% of rectal polyps >3cm contain a malignant component. Similarly, in recent studies it was shown that 10-15% of entirely benign polyps were removed by abdominal surgery rather than endoscopically. This has major implications for the patient since surgical resection is associated with considerable morbidity. Therefore, there is a need of a technique that provide the endoscopist with real-time information about specific molecular features of the tumor to differentiate between benign polyps with LGD amenable for pEMR and those that contain HGD or T1RC that require en-bloc resection. Tumor targeted fluorescence-guided surgery (FGS) has emerged as a technique with the potential to enable real-time lesion visualization based on specific molecular features rather than on morphology. Recently it was shown that carcinoembryonic antigen (CEA) is overexpressed in approximately 75% of T1RC/HGD. Additionally, expression in LGD was (nearly) absent in 66% of low-grade dysplastic tissue and in 98% of normal rectum tissue, making it a suitable marker for distinguishing T1RC and HGD from LGD and normal tissue. CEA can be targeted by SGM-101, an anti-CEA antibody attached to a fluorophore which has been studied in several clinical studies for patients with colorectal cancer undergoing surgery. The investigators hypothesize that the use of SGM-101 during endoscopy aids the endoscopist in discriminating benign polyps with solely LGD from polyps containing T1RC/HGD.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have suspected T1RC/HGD and scheduled for a local endoscopic en-bloc resection. The rectum is defined as the area between the linea dentata and 10cm ab ano.
2. Age > 18 years old
3. Patients should be capable and willing to give signed informed consent before study specific procedures.

Exclusion Criteria:

1. Prior participation in this study
2. Previous administration of SGM-101
3. Patients with a history of anaphylactic shock
4. Patients pregnant or breastfeeding, lack of effective contraception in male or female patients with reproductive potential
5. Any condition that the investigator considers to be potentially jeopardizing the patients' well-being or the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
The ex-vivo NIR-fluorescence tumour to dysplasia ratio (TDR, T1RC/HGD to LGD ratio) on bread loafs (macroscopic) and pathology slides (microscopic). | 1.5 years
  The ex-vivo NIR-fluorescence tumour to dysplasia ratio (TDR, T1RC/HGD to LGD ratio) on bread loafs (macroscopic) and pathology slides (microscopic).

SECONDARY OUTCOMES:
- Ex-vivo NIR-fluorescence tumour-to-background ratio (TBR) and dysplasia-to-background ratio (DBR) (ex-vivo TDR already encountered within main objective) | 1.5 years
- In-vivo TDR, TBR and DBR, as measured with the Quest spectrum laparoscope. | 1.5 years
- The accuracy of SGM-101 to discriminate T1RC/HGD from LGD ex-vivo | 1.5 years
-The accuracy of SGM-101 to discriminate T1RC/HGD from LGD in-vivo | 1.5 years
- The correlation between in-vivo TBR/TDR and Kudo level (SM1 vs SM2/3) | 1.5 years
- The agreement of resection margins status (R0 vs R1) assessed by fluorescence and histopathology. A resection margin is classified positive when there is a fluorescent hotspot visible in the wound bed or on the specimen. | 1.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data will be coded and available only to the researchers of the LUMC on this particular trial. No other people will get access to the data. Results will be published.